CLINICAL TRIAL: NCT02542176
Title: Pilot Study: Effects of a Standardized Freeze-dried Grape Powder on High Density Lipoprotein (HDL) Function in Metabolic Syndrome
Brief Title: Effects of a Standardized Freeze-dried Grape Powder on High Density Lipoprotein (HDL) Function in Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Collaborators: California Table Grape Commission (Other)
Responsible Party: Principal Investigator, Christopher Blesso, Assistant Professor, University of Connecticut
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 150888
Record Dates: First submitted 2015-09-01; First posted 2015-09-04 (Estimated); Last update posted 2018-03-23 (Actual); Status verified 2018-03

CONDITIONS: Metabolic Syndrome X
Keywords: Metabolic Syndrome; Grape; HDL; Lipoproteins
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Freeze-dried Whole Grape Powder (Experimental)
  Interventions: Other: Freeze-dried Whole Grape Powder
- Grape Powder Placebo (Placebo Comparator)
  Interventions: Other: Grape Powder Placebo

INTERVENTIONS:
Other: Freeze-dried Whole Grape Powder — 60 g of whole grape powder for 4 weeks
  Arms: Freeze-dried Whole Grape Powder
Other: Grape Powder Placebo — 60 g of grape powder placebo for 4 weeks
  Arms: Grape Powder Placebo

SUMMARY:
The purpose of this study is to evaluate the effects of both chronic and acute grape ingestion in a population of men and women at higher risk for both type 2 diabetes and cardiovascular disease (metabolic syndrome).

DETAILED DESCRIPTION:
This study will involve a 2-week "run-in" period and two 4-week "intervention" phases separated by a 3 week "washout" non-intervention phase (for a total of 13 weeks). At the start of each 4-week intervention period, subjects will be asked to participate in a "postprandial challenge" test. Subjects will be asked to first follow a 2-week run-in control period consuming habitual diets but refraining from consuming polyphenol-rich foods/beverages, including tea, berries, grapes, juices, and wine. Subjects will then be asked to consume 60 g of grape powder or placebo in random order, each for a 4-week intervention period, separated by a 3-week washout period. Subjects will be asked to prepare powder by mixing with water at breakfast (30 g) and dinner (30 g) and consume immediately after mixing (or within 30 minutes). During each 4-week intervention period, subjects will be asked to refrain from consuming polyphenol-rich foods/beverages. During the washout period subjects will not be asked to consume the powder, but should abstain from consuming polyphenol-rich foods/beverages. The grape powder is made from a composite of fresh red, green and black California grapes, based on actual consumption patterns of consumers. It is a mix of seeded and seedless varieties that have been frozen, ground with food-quality dry ice, freeze-dried, and re-ground. Subjects will also be asked to maintain normal diet and exercise habits throughout the study, with the exception being the consumption of polyphenol-rich foods/beverages. Subjects will be asked to complete a 5-day dietary record (including 1 weekend day) and a 7-day physical activity diary at the baseline and end of each intervention period. Subjects will come to the University of Connecticut Nutrition Department once every other week (biweekly) to pick up the powder (in packets), which needs to be kept frozen until consumption.

For the postprandial challenge tests, subjects will be asked to fast overnight (12 hours) and then will be given a coconut oil-based lactose-free milkshake (1 g fat/kg body weight), containing 60 g of either placebo or grape powder. Subjects will be asked to spend the test day in the laboratory in a rested state and, with the exception of water, will not be permitted to consume any additional food or beverages during the 6 hours after consuming the milkshake. Subjects will be asked to abstain from alcohol and strenuous physical activity 24-hours prior to the postprandial test. To standardize short-term fat intake, subjects will be given recipes and instructed to consume a low-fat evening meal (< 10 g fat) the night prior to postprandial tests. Subjects will also be asked to complete a 1-day food record for the day prior to the postprandial tests.

ELIGIBILITY:
Inclusion Criteria:

* Age 30 to 70 years
* Having metabolic syndrome, meaning that subjects have at least 3 of the following characteristics:
* Waist circumference ≥ 102 cm for men and ≥ 88 cm for women
* Triglycerides ≥ 150 mg/dL
* HDL cholesterol < 40 mg/dL for men and < 50 mg/dL for women
* Blood pressure ≥ 130/85 mm Hg or taking an anti-hypertensive medication
* Fasting blood glucose ≥ 100 mg/dL

Exclusion Criteria:

* Do not fulfill the classification of metabolic syndrome
* History of diabetes mellitus, cardiovascular disease, stroke, renal problems, liver disease, endocrine disorder, inborn error of metabolism, eating disorder or cancer.
* Weight loss greater than 10% of body weight over preceding 4 weeks.
* Taking high-dose aspirin (≥150 mg/day) or anti-inflammatory prescriptions, or any triglyceride- or glucose-lowering prescriptions or supplements, such as insulin, sodium-glucose transport protein-2 (SGLT-2) inhibitors, glucagon-like peptide-1 (GLP-1) agonists, Fibrates (e.g., fenofibrates, gemfibrozil), Niacin (e.g., high dose nicotinic acid, Niaspan) Sulphonylureas (e.g., Glucotrol, Amaryl), Thiazolidinediones (e.g., Avandia, ACTOS, Rezulin), Meglitinides (e.g., Prandin, Starlix), Biguanides (e.g., Metformin), Alpha-glucosidase inhibitors (e.g., Precose, Glyset), dipeptidyl peptidase-4 (DPP-4) inhibitors (e.g., Januvia, Onglyza), prescription fish oil (e.g., Lovaza, Vascepa), high dose chromium, high dose fish oil, or cinnamon supplements etc.
* Triglycerides are higher than 500 mg/dL, glucose levels higher than 126 mg/dL, blood pressure higher than 160/100 mmHg, and waist circumference higher than 200 cm.
* Allergy to coconut, milk, wheat, grapes or an allergy/intolerance to the placebo ingredients.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-10; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Fasted HDL-cholesterol | 13 weeks
  Measurement of plasma HDL-cholesterol (mg/dL) at the end of each 4-week intervention arms.

SECONDARY OUTCOMES:
Fasted apolipoprotein B-depleted serum cholesterol efflux capacity | 13 weeks
  Measurement of fasted apolipoprotein B-depleted serum cholesterol efflux capacity (% cholesterol efflux) from macrophages loaded with tritium(3H)-labeled-cholesterol at the end of each 4-week intervention arms. Results will be expressed as percent efflux calculated as disintegrations per minute of [3H]-cholesterol in medium ÷ ([3H]-cholesterol in medium + [3H]-cholesterol remaining in cells) x 100.
Postprandial HDL anti-inflammatory activity | On first day of each intervention arm up to 6 hours after test meal
  Adhesion molecule expression (micrograms/L) will be measured after incubation of human endothelial cells with HDL isolated from pre-test meal (baseline), 3 hours post-test meal, and 6 hours post-test meal time points.
Postprandial HDL antioxidant activity | On first day of each intervention arm up to 6 hours after test meal
  Paraoxonase-1 enzyme activity towards phenyl acetate (kU/L) measured in serum from pre-test meal (baseline), 3 hours post-test meal, and 6 hours post-test meal time points.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Connecticut, Storrs, Connecticut, United States

REFERENCES:
- [Derived] Millar CL, Duclos Q, Garcia C, Norris GH, Lemos BS, DiMarco DM, Fernandez ML, Blesso CN. Effects of Freeze-Dried Grape Powder on High-Density Lipoprotein Function in Adults with Metabolic Syndrome: A Randomized Controlled Pilot Study. Metab Syndr Relat Disord. 2018 Nov;16(9):464-469. doi: 10.1089/met.2018.0052. Epub 2018 Aug 21. PMID 30129815